**Title:** PRMRP Norms: Iterative Design of Custom Dynamic Orthoses and Comprehensive Design of Musculoskeletal Model.

NCT Number: NCT04800510

Date: November 7, 2023

## **Study Protocol:**

# Purpose and Procedures:

The purpose of this study is to determine the effect of external bracing, in the form of a carbon fiber dynamic orthosis, on joint contact stress, muscle forces, physical function, and gait biomechanics. The effects of external bracing on gait mechanics, mobility, and muscle and joint forces are poorly understood. Collected data will include patient demographics and anthropometrics, ankle range of motion and stiffness data, plantarflexion strength data, CT images, CDO stiffness data, physical performance measures, patient reported outcomes, gait kinematics and kinetics, plantar pressures, and electromyography data. The knowledge that will be gained from this investigation has the potential to substantially improve the understanding of how external bracing impacts limb function and inform future investigations to advance the clinical prescription of ankle foot orthoses.

# Objectives and Specific Aims:

Specific Aim 1: Determine the effect of CDO design modifications on ankle contact stress in a cohort of healthy able-bodied individuals.

Specific Aim 2: Determine the effect of CDO design modifications on physical function and gait biomechanics in a cohort of healthy able-bodied individuals.

Specific Aim 3: Determine the effect of CDO design modification on muscle forces during gait

Specific Aim 4: Refine methods of integrating data from multiple sources into musculoskeletal model to evaluate ankle contact stress.

# Background and Significance:

Post-traumatic osteo-arthritis (PTOA) is a significant problem caused by chronic, increased, contact stress and fracture severity. Surgical fracture reduction has been the mainstay of intra-articular fracture (IAF) treatment for decades, but it is not the only factor influencing joint contact stresses. Furthermore, even with the best surgical effort, there often remains residual incongruity that leads to elevated contact stress. Numerous studies have explored the relationship between elevated contact stresses and the development of osteoarthritis following traumatic injury of the ankle. CDOs, such as the Intrepid Dynamic Exoskeletal Orthosis (IDEO) developed at Brooke Army Medical Center, have been used to dramatically improve function and reduce pain in hundreds of service members with traumatic limb injury. CDOs are comprised of a proximal cuff sitting just below the knee, a posterior strut used to store and return energy, a semi-rigid foot plate, and in some cases a heel cushion between the footplate and shoe [11]. These design components can be varied to influence the forces and motions experienced by the limb [11-14], which in turn influence the forces on the foot and the activation of muscles that cross the ankle [8, 15, 16]. Recent findings indicate that this can decrease load transfer across the ankle, which implies that CDOs may be able to be effectively tuned to reduce articular contact stress. A key mechanism by which may articular contact stress may be reduced is the reduction of force produced by muscles around the ankle.

The multiple data sources collected in this study will serve as inputs for creating a comprehensive musculoskeletal model using OpenSim modeling software. OpenSim is an extensible software package that has been developed over decades to combine knowledge of computational modeling and biomechanical system simulations in order to calculate muscle forces generated from movement, kinematic adaptations during gait, and human-device interactions [78]. The use of OpenSim will allow for accurate simulations of gait, as well as calculation and prediction of variables that are difficult to measure experimentally [78].

## Inclusion/Exclusion Criteria:

#### Patient Inclusion Criteria

- Between the ages of 18 and 50
- Shoe size between women's 8 and 13.5 or men's 6.5 and 12
- Healthy individuals without a current complaint of lower extremity pain, spine pain, or medical

or neuromusculoskeletal disorders that have limited participation in work or exercise in the last 6 months

- Full active range of motion of the bilateral lower extremities and spine
- Ability to hop without pain
- Ability to perform a full squat without pain
- Ability to read and write in English and provide written informed consent

## Patient Exclusion Criteria

- Diagnosed moderate or severe brain injury
- Prior lower extremity injury resulting in surgery or limiting function for greater than 6 weeks
- Diagnosis of a physical or psychological condition that would preclude testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
- Visual or hearing impairment that would interfere with instructions given during testing
- Require an assistive device
- Wounds to the foot or calf that would prevent CDO use
- BMI greater than 35
- Pregnancy Per participant self-report. Due to the expected small number of pregnant individuals and resulting inability to account for its effect on resulting outcomes, participants will be withdrawn from the study

#### Design and Methods:

Patients will wear generic sized CDOs provided by Bio-Mechanical Composites (Des Moines, IA). Personal/demographic and anthropometric information will be used to fully characterize the study participants. We will collect multiple variables that have been previously associated with outcomes including race, ethnicity, and education. Anthropometric and demographic information such as age, biological sex, study limb (left or right), height, weight, leg length, shoe type, shoe length and width will also be used to characterize the cohort. Multiple outcomes measures will be used to characterize patient-centric outcomes.

Physical performance measures provide an objective and responsive assessment of an individual's functional mobility. Activities of daily life require performance of a range of functional tasks that require balance, agility, speed, and power. The four square step test (4SST) is a widely used test of functional mobility that requires rapid changes in direction that are often problematic following lower limb injury. The measure has good to excellent reliability and validity across multiple patient populations and groups and is a key dependent measure in most CDO-related studies to date and has demonstrated ability to detect changes in function in individuals with limb trauma and CDOs [7, 9, 27, 36]. The sit to stand 5 times (STS5) test is a well-established measure of lower limb muscle strength, endurance, and mobility [39]. The STS5 test has excellent reliability and good validity across a broad range of patient populations [35, 39-48].

Patient-reported outcomes questionnaires will be used to evaluate participant physical function, activity level, pain, comfort, satisfaction, and preference in addition to multiple other relevant outcomes. The Orthotics Prosthetics Users' Survey (OPUS) is a leading measure for evaluating satisfaction with orthotic devices and services [49]. It is a self-report questionnaire, with the full battery consisting of 88 questions and five modules. The satisfaction with devices portion will be used to evaluate device comfort, form, and fit using a four-point Likert scale and has good to excellent reliability, internal consistency, and validity for individuals with a wide range of diagnoses requiring orthotic and prosthetic services [49]. Comfort and smoothness will also be assessed using a modified version of the Socket Comfort Score, a reliable, valid, and sensitive measure of device fit and comfort [50]. These measures have been shown to effectively capture patient perception, are

responsive to simple modifications to CDO device function, and will be applied in a manner consistent with a prior publication by the research team [11]. Participants will be asked to report their pain using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable, at the start of each session, and at multiple points while walking in each condition. Participants will be asked to rate the three braces (CDO-A, CDO-B, and CDO-C) on a standard 11-point scale, where 0 = worst imaginable device and 10 = best imaginable device. The University of California, Los Angeles (UCLA) activity score is a 10-level rating scale that is used to both qualitatively and quantitatively define an individual's current and/or desired level of activity and has been shown to be reliable with no floor effects [53]. The Patient Reported Outcomes Measurement Information System (PROMIS) is a group of patient-centered tests, developed through funding from the National Institutes of Health, which can be used to characterize physical, mental, and social health and function. The PROMIS instruments use modern measurement theory to reliably and validly assess patient-reported outcomes. We will use PROMIS to evaluate physical function. Semi-structured interviews will also be used to fully capture the patients' perspectives, experience, and opinions associated with the device options they experienced as part of the study.

Impairment, biomechanical, and device data will be used to compare devices, characterize limb and device function, and to provide insight in a manner not commonly found in comparative studies. Bending stiffness will be measured using a custom-made orthotic stiffness testing device designed specifically for quantifying CDO bending stiffness in Nm/degree. Ground reaction force and motion capture data will be used to evaluate the motion and loading of the lower limb and CDO devices as participants walk on an over ground walkway at self-selected speed and a controlled speed based on leg length [54, 55]. Muscle activity will be measured using DELSYS EMG sensors. EMG data will be collected bilaterally in the lower limbs and data will be analyzed over regions throughout the gait cycle. In-shoe plantar pressure distribution will be measured using the LoadSol system which interfaces with the foot and shoe insole and has been found to be accurate, precise, and repeatable in measuring plantar pressures during normal gait [60, 61]. Ankle range of motion and stiffness will be assessed using the Iowa Ankle Range of Motion device. Ankle strength will be assessed using the Standing Heel-Rise Test. Subjects will perform as many standing heel-rises as they can, while their ankle motion and body/limb alignment are carefully monitored.

#### **Statistical Analysis Plan:**

#### Analysis Methods:

Data quality will be rigorously examined over the course of this study. The distributions of study measures will be characterized using descriptive statistics. For descriptive statistics, univariate statistical approaches will include careful review of data frequencies, measures of central tendency, and distribution shapes. Additionally, identification of out of range data, determination of the quantity of missing data, and accurate description of the study population will be achieved.

## Power Analysis:

The proposed sample size for this study is 10 subjects. Since the primary purpose of this study is to refine procedures for inputting multiple data sources into a musculoskeletal model, the study does not call for a total number of participants consistent with prior investigations by Dr. Wilken. In a 2017 study conducted by Blazkiewicz et al, data was collected from 10 healthy subjects and incorporated into a generic OpenSim musculoskeletal model [79]. The results of the study showed some inter-individual variation as expected, but identified a common theme of muscle peak force regularities acting on the ankle joint across subjects, indicating that a 10 subject sample size is sufficient for the protocol design of similar investigations [79].

## **References Cited:**

- 1. Anderson, D.D., et al., Intra-articular contact stress distributions at the ankle throughout stance phase-patient-specific finite element analysis as a metric of degeneration propensity. Biomech Model Mechanobiol, 2006. 5(2-3): p. 82-9.
- 2. Anderson, D.D., J.L. Marsh, and T.D. Brown, The pathomechanical etiology of post-traumatic osteoarthritis following intraarticular fractures. Iowa Orthop J, 2011. 31: p. 1-20.
- 3. Kern, A.M. and D.D. Anderson, Expedited patient-specific assessment of contact stress exposure in the ankle joint following definitive articular fracture reduction. J Biomech, 2015. 48(12): p. 3427-32.
- 4. Anderson, D.D., et al., Expedited CT-Based Methods for Evaluating Fracture Severity to Assess Risk of Post-Traumatic Osteoarthritis After Articular Fractures. Iowa Orthop J, 2016. 36: p. 46-52.
- 5. Anderson, D.D., et al., Is elevated contact stress predictive of post-traumatic osteoarthritis for imprecisely reduced tibial plafond fractures? J Orthop Res, 2011. 29(1): p. 33-9.
- 6. Amorelli, C.R., et al., Center for the Intrepid: Providing Patients POWER. US Army Med Dep J, 2016: p. 39-46.
- 7. Bedigrew, K.M., et al., Can an integrated orthotic and rehabilitation program decrease pain and improve function after lower extremity trauma? Clin Orthop Relat Res, 2014. 472(10): p. 3017-25.
- 8. Brown, S.E., E. Russell Esposito, and J.M. Wilken, The effect of ankle foot orthosis alignment on walking in individuals treated for traumatic lower extremity injuries. J Biomech, 2017. 61: p. 51-57.
- 9. Hsu, J.R., et al., Patient Response to an Integrated Orthotic and Rehabilitation Initiative for Traumatic Injuries: The PRIORITI-MTF Study. J Orthop Trauma, 2017. 31 Suppl 1: p. S56-S62.
- 10. Russell Esposito, E., et al., Gait biomechanics following lower extremity trauma: Amputation vs. reconstruction. Gait Posture, 2017. 54: p. 167-173.
- 11. Ikeda, A.J., J.R. Fergason, and J.M. Wilken, Effects of altering heel wedge properties on gait with the Intrepid Dynamic Exoskeletal Orthosis. Prosthet Orthot Int, 2018. 42(3): p. 265-274.
- 12. Haight, D.J., E. Russell Esposito, and J.M. Wilken, Biomechanics of uphill walking using custom ankle-foot orthoses of three different stiffnesses. Gait Posture, 2015. 41(3): p. 750-6.
- 13. Russell Esposito, E., et al., How does ankle-foot orthosis stiffness affect gait in patients with lower limb salvage? Clin Orthop Relat Res, 2014. 472(10): p. 3026-35.
- 14. Russell Esposito, E., et al., Biomechanical response to ankle-foot orthosis stiffness during running. Clin Biomech (Bristol, Avon), 2015. 30(10): p. 1125-32.
- 15. Harper, N.G., et al., The influence of ankle-foot orthosis stiffness on walking performance in individuals with lower-limb impairments. Clin Biomech (Bristol, Avon), 2014. 29(8): p. 877-84.
- 16. Ranz, E.C., et al., The influence of passive-dynamic ankle-foot orthosis bending axis location on gait performance in individuals with lower-limb impairments. Clin Biomech (Bristol, Avon), 2016. 37: p. 13-21.
- 17. Hancock, K., et al., Efficacy of Multimodal Analgesic Injections in Operatively Treated Ankle Fractures: A Randomized Controlled Trial. The Journal of Bone and Joint Surgery, 2019. 101: p. 1.
- 18. Plumarom, Y., et al., Radiographic Healing of Far Cortical Locking Constructs in Distal Femur Fractures: A Comparative Study with Standard Locking Plates. Journal of Orthopaedic Trauma, 2019: p. 1.
- 19. Kern, A.M., et al., Intra-OP biomechanical guidance improves articular fracture reduction, limiting post-traumatic OA risk. Osteoarthritis and Cartilage, 2018. 26: p. S375.
- 20. Coleman, M., et al., Targeting mitochondrial responses to intra-articular fracture to prevent posttraumatic osteoarthritis. Science Translational Medicine, 2018. 10: p. eaan5372.

- 21. Coleman, M., et al., Intraarticular Administration of N-Acetylcysteine Prevents Progression of Post-Traumatic Osteoarthritis in a Large Animal Model of Intraarticular Fracture. Free Radical Biology and Medicine, 2015. 87: p. S88-S89.
- 22. Barg, A., et al., Weightbearing Computed Tomography of the Foot and Ankle: Emerging Technology Topical Review. Foot Ankle Int, 2018. 39(3): p. 376-386.
- 23. Lintz, F., et al., Weight-bearing cone beam CT scans in the foot and ankle. EFORT Open Rev, 2018. 3(5): p. 278-286.
- 24. Russell Esposito, E., et al., Ankle-foot orthosis bending axis influences running mechanics. Gait Posture, 2017. 56: p. 147-152.
- 25. Aldridge Whitehead, J.M., E. Russell Esposito, and J.M. Wilken, Stair ascent and descent biomechanical adaptations while using a custom ankle-foot orthosis. J Biomech, 2016. 49(13): p. 2899-2908.
- 26. Patzkowski, J.C., et al., Can an ankle-foot orthosis change hearts and minds? J Surg Orthop Adv, 2011. 20(1): p. 8-18.
- 27. Patzkowski, J.C., et al., Comparative effect of orthosis design on functional performance. J Bone Joint Surg Am, 2012. 94(6): p. 507-15.
- 28. Sheean, A.J., et al., Effect of Custom Orthosis and Rehabilitation Program on Outcomes Following Ankle and Subtalar Fusions. Foot Ankle Int, 2016. 37(11): p. 1205-1210.
- 29. Aldridge, J.M., J.T. Sturdy, and J.M. Wilken, Stair ascent kinematics and kinetics with a powered lower leg system following transtibial amputation. Gait Posture, 2012. 36(2): p. 291-5.
- 30. Harper, N.G., et al., Selective laser sintered versus carbon fiber passive-dynamic ankle-foot orthoses: a comparison of patient walking performance. J Biomech Eng, 2014. 136(9): p. 091001.
- 31. O'Toole, R.V., et al., Determinants of patient satisfaction after severe lower-extremity injuries. J Bone Joint Surg Am, 2008. 90(6): p. 1206-11.
- 32. Archer, K.R., et al., Physical disability after severe lower-extremity injury. Arch Phys Med Rehabil, 2006. 87(8): p. 1153-5.
- 33. MacKenzie, E.J., et al., Characterization of patients with high-energy lower extremity trauma. J Orthop Trauma, 2000. 14(7): p. 455-66.
- 34. Doukas, W.C., et al., The Military Extremity Trauma Amputation/Limb Salvage (METALS) study: outcomes of amputation versus limb salvage following major lower-extremity trauma. J Bone Joint Surg Am, 2013. 95(2): p. 138-45.
- 35. Wilken, J.M., et al., Physical performance assessment in military service members. J Am Acad Orthop Surg, 2012. 20 Suppl 1: p. S42-7.
- 36. Dite, W. and V.A. Temple, A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil, 2002. 83(11): p. 1566-71.
- 37. Whitney, S.L., et al., The reliability and validity of the Four Square Step Test for people with balance deficits secondary to a vestibular disorder. Arch Phys Med Rehabil, 2007. 88(1): p. 99-104.
- 38. Dite, W., H.J. Connor, and H.C. Curtis, Clinical identification of multiple fall risk early after unilateral transtibial amputation. Arch Phys Med Rehabil, 2007. 88(1): p. 109-14.
- 39. Whitney, S.L., et al., Clinical measurement of sit-to-stand performance in people with balance disorders: validity of data for the Five-Times-Sit-to-Stand Test. Phys Ther, 2005. 85(10): p. 1034-45.
- 40. Wang, T.H., H.F. Liao, and Y.C. Peng, Reliability and validity of the five-repetition sit-to-stand test for children with cerebral palsy. Clin Rehabil, 2012. 26(7): p. 664-71.

- 41. Paul, S.S., et al., Reproducibility of measures of leg muscle power, leg muscle strength, postural sway and mobility in people with Parkinson's disease. Gait Posture, 2012. 36(3): p. 639-42.
- 42. Mong, Y., T.W. Teo, and S.S. Ng, 5-repetition sit-to-stand test in subjects with chronic stroke: reliability and validity. Arch Phys Med Rehabil, 2010. 91(3): p. 407-13.
- 43. Lin, Y.C., R.C. Davey, and T. Cochrane, Tests for physical function of the elderly with knee and hip osteoarthritis. Scand J Med Sci Sports, 2001. 11(5): p. 280-6.
- 44. Bohannon, R.W., Reference values for the five-repetition sit-to-stand test: a descriptive meta-analysis of data from elders. Percept Mot Skills, 2006. 103(1): p. 215-22.
- 45. Duncan, R.P., A.L. Leddy, and G.M. Earhart, Five times sit-to-stand test performance in Parkinson's disease. Arch Phys Med Rehabil, 2011. 92(9): p. 1431-6.
- 46. Beninato, M., L.G. Portney, and P.E. Sullivan, Using the International Classification of Functioning, Disability and Health as a framework to examine the association between falls and clinical assessment tools in people with stroke. Phys Ther, 2009. 89(8): p. 816-25.
- 47. Newcomer, K.L., H.E. Krug, and M.L. Mahowald, Validity and reliability of the timed-stands test for patients with rheumatoid arthritis and other chronic diseases. J Rheumatol, 1993. 20(1): p. 21-7.
- 48. Schaubert, K.L. and R.W. Bohannon, Reliability and validity of three strength measures obtained from community-dwelling elderly persons. J Strength Cond Res, 2005. 19(3): p. 717-20.
- 49. Peaco, A., Halsne E., Hafner, BJ., Assessing Satisfaction With Orthotic Devices and Services: A Systematic Literature Review. Journal of Prosthetics and Orthotics, 2011. 23(2): p. 95-105.
- 50. Hanspal, R.S., K. Fisher, and R. Nieveen, Prosthetic socket fit comfort score. Disabil Rehabil, 2003. 25(22): p. 1278-80.
- 51. Hjermstad, M.J., et al., Studies comparing Numerical Rating Scales, Verbal Rating Scales, and Visual Analogue Scales for assessment of pain intensity in adults: a systematic literature review. J Pain Symptom Manage, 2011. 41(6): p. 1073-93.
- 52. Williamson, A. and B. Hoggart, Pain: a review of three commonly used pain rating scales. J Clin Nurs, 2005. 14(7): p. 798-804.
- 53. Naal, F.D., F.M. Impellizzeri, and M. Leunig, Which is the best activity rating scale for patients undergoing total joint arthroplasty? Clin Orthop Relat Res, 2009. 467(4): p. 958-65.
- 54. Wilken, J.M., et al., Reliability and Minimal Detectible Change values for gait kinematics and kinetics in healthy adults. Gait Posture, 2012. 35(2): p. 301-7.
- 55. Vaughan, C.L. and M.J. O'Malley, Froude and the contribution of naval architecture to our understanding of bipedal locomotion. Gait Posture, 2005. 21(3): p. 350-62.
- 56. Kaufman, K., et al., Reliability of 3D gait data across multiple laboratories. Gait Posture, 2016. 49: p. 375-381.
- 57. De Asha, A.R., et al., Attenuation of centre-of-pressure trajectory fluctuations under the prosthetic foot when using an articulating hydraulic ankle attachment compared to fixed attachment. Clin Biomech (Bristol, Avon), 2013. 28(2): p. 218-24.
- 58. De Asha, A.R., et al., Impact on the biomechanics of overground gait of using an 'Echelon' hydraulic anklefoot device in unilateral trans-tibial and trans-femoral amputees. Clin Biomech (Bristol, Avon), 2014. 29(7): p. 728-34.
- 59. Klenow, T.D., J.T. Kahle, and M.J. Highsmith, The dead spot phenomenon in prosthetic gait: Quantified with an analysis of center of pressure progression and its velocity in the sagittal plane. Clin Biomech (Bristol, Avon), 2016. 38: p. 56-62.

- 60. Hsiao, H., J. Guan, and M. Weatherly, Accuracy and precision of two in-shoe pressure measurement systems. Ergonomics, 2002. 45(8): p. 537-55.
- 61. Ramanathan, A.K., et al., Repeatability of the Pedar-X in-shoe pressure measuring system. Foot Ankle Surg, 2010. 16(2): p. 70-3.
- 62. Wilken, J., et al., A new device for assessing ankle dorsiflexion motion: reliability and validity. J Orthop Sports Phys Ther, 2011. 41(4): p. 274-80.
- 63. Archer, K.R., et al., Gait symmetry and walking speed analysis following lower-extremity trauma. Phys Ther, 2006. 86(12): p. 1630-40.
- 64. Castillo, R.C., et al., Evidence of beneficial effect of physical therapy after lower-extremity trauma. Arch Phys Med Rehabil, 2008. 89(10): p. 1873-9.
- 65. Hancock, M.J., R.D. Herbert, and M. Stewart, Prediction of outcome after ankle fracture. J Orthop Sports Phys Ther, 2005. 35(12): p. 786-92.
- 66. Burns, J. and J. Crosbie, Weight bearing ankle dorsiflexion range of motion in idiopathic pes cavus compared to normal and pes planus feet. The Foot, 2005. 15(2): p. 91-94.
- 67. Konor, M.M., et al., Reliability of three measures of ankle dorsiflexion range of motion. Int J Sports Phys Ther, 2012. 7(3): p. 279-87.
- 68. Hicks, J.H., The mechanics of the foot. I. The joints. J Anat, 1953. 87(4): p. 345-57.
- 69. Ikeda AJ, Fergason JR, Wilken JM. Clinical Outcomes with the Intrepid Dynamic Exoskeletal Orthosis: A Retrospective Analysis. Mil Med. 2019;184(11-12):601‐605. doi:10.1093/milmed/usz004
- 70. Anderson, D.D., et al., Physical validation of a patient-specific contact finite element model of the ankle. J Biomech, 2007. 40(8): p. 1662-9.
- 71. Fitzpatrick, D.C., et al., Kinematic and contact stress analysis of posterior malleolus fractures of the ankle. J Orthop Trauma, 2004. 18(5): p. 271-8.
- 72. Haraguchi, N., et al., Prediction of three-dimensional contact stress and ligament tension in the ankle during stance determined from computational modeling. Foot Ankle Int, 2009. 30(2): p. 177-85.
- 73. Kraeutler, M.J., et al., Peculiarities in Ankle Cartilage. Cartilage, 2017. 8(1): p. 12-18.
- 74. McKinley, T.O., et al., Instability-associated changes in contact stress and contact stress rates near a step-off incongruity. J Bone Joint Surg Am, 2008. 90(2): p. 375-83.
- 75. Liu, Q., et al., Analysis of the stress and displacement distribution of inferior tibiofibular syndesmosis injuries repaired with screw fixation: a finite element study. PLoS One, 2013. 8(12): p. e80236.
- 76. Guan, M., et al., Finite element analysis of the effect of sagittal angle on ankle joint stability in posterior malleolus fracture: A cohort study. Int J Surg, 2019. 70: p. 53-59.
- 77. Lintz, F., et al., Weight-bearing cone beam CT scans in the foot and ankle. EFORT Open Rev, 2018. 3(5): p. 278-286.
- 78. Seth, A., et al., OpenSim: Simulating musculoskeletal dynamics and neuromuscular control to study human and animal movement. PLoS Comput Biol, 2018. 14(7): p. e1006223.
- 79. Blazkiewicz, M., et al., Inter-individual similarities and variations in muscle forces acting on the ankle joint during gait. Gait Posture, 2017. 58: p. 166-170